CLINICAL TRIAL: NCT02134067
Title: A Phase 1, Open-Label, Non-Randomized, Dose-Escalating Safety, Tolerability and Pharmacokinetic Study of TAS-119 in Combination With Paclitaxel in Patients With Advanced Solid Tumors
Brief Title: Dose-escalating, Safety, Tolerability and PK Study of TAS-119 in Combination With Paclitaxel in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TO-TAS-119-101
Record Dates: First submitted 2014-04-28; First posted 2014-05-08 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumors
Keywords: advanced solid tumors; tumor; Dose Escalation; TAS-119; Taxane; Paclitaxel; Aurora A kinase inhibitor; AurA
MeSH Terms: conditions — Neoplasms; Epilepsy | interventions — TAS-119; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAS-119 (Experimental): TAS-119 tablets, oral, dose-escalating, 28-day cycle.
  Paclitaxel (90mg/m2) is administered IV in combination with TAS-119 in each of the arms.
  Interventions: Drug: TAS-119; Drug: Paclitaxel

INTERVENTIONS:
Drug: TAS-119
Drug: Paclitaxel — A dose of 90 mg/m2 is used in combination with various doses of TAS-119.
  Other Names: Taxol

SUMMARY:
The purpose of this study is to determine the safety of TAS-119 and determine the most appropriate dose in combination with Paclitaxel for subsequent studies in patients with advanced solid tumors.

TAS-119 is a novel, selective Aurora A kinase inhibitor, which has previously been demonstrated to enhance the activity of paclitaxel in preclinical studies

DETAILED DESCRIPTION:
Background and rationale for study:

In nonclinical pharmacology studies TAS-119 significantly enhanced the antitumor activity of the microtubule stabilizer paclitaxel and TAS-119 is being developed for use in combination with paclitaxel.

TAS-119 selectively inhibits the kinase inhibitor Aurora A. AurA regulates cell division by controlling the transition from G2 to M phase. Overexpression of AurA is associated with resistance to taxanes.

The study will be conducted in two sequential phases:

Dose Escalation Phase with the purpose to determine the maximum tolerated dose and the recommended Phase 2 dose of TAS-119 given in combination with paclitaxel

An Expansion Phase in which additional patients will be enrolled to further evaluate the safety and preliminary efficacy of the recommended Phase 2 dose of TAS-119 in combination with paclitaxel, during which a subgroup of patients will be evaluated for DDI between paclitaxel and TAS-119 via PK assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or female ≥ 18 years of age, that has provided written informed consent.
2. Has histologically or cytologically confirmed advanced, unresectable metastatic solid tumor(s) for which the patients have no available therapy likely to provide clinical benefit, or for which paclitaxel is considered a standard of care.
3. Has adequate organ function as defined by the following criteria:

   * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 3.0 × upper limit of normal (ULN); if liver function abnormalities are due to underlying liver metastasis, AST (SGOT) and ALT (SGPT) ≤ 5 × ULN.
   * Total serum bilirubin ≤ 1.5 × ULN.
   * Absolute neutrophil count ≥ 1,500/mm3 (excluding measurements obtained within 7 days after administration of granulocyte colony-stimulating factor [G-CSF]).
   * Platelet count ≥ 100,000/mm3 (IU: ≥ 100 × 109/L) (excluding measurements obtained within 7 days after a transfusion of platelets).
   * Hemoglobin ≥ 9.0 g/dL
   * Total serum creatinine ≤ 1.5 × ULN
   * Serum albumin ≥ 3.0 mg/dL.

Exclusion Criteria:

1. Previous inability to tolerate any dose of paclitaxel (i.e., the subject required a paclitaxel dose reduction or discontinuation).
2. Has received any treatments prohibited in this trial within specified time frames
3. Has a serious illness or medical condition(s) that would affect safety or tolerability of the study treatments
4. Has history of Grade 2 or greater peripheral neuropathy during the 3 months prior to enrollment.
5. Has known hypersensitivity to TAS-119 or its components.
6. Has known hypersensitivity to Cremophor® EL, paclitaxel or its components.
7. Is a pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of TAS-119 in combination with paclitaxel | Safety monitoring will begin at the time of the first dose of TAS-119, and will continue until all patients are discontinued from treatment or until 12 months from the last patient enrolled (up to 3 years).
  Standard safety monitoring and grading using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 will be used.
  The safety and tolerability of TAS-119 will be evaluated by the number and severity of adverse events, vital signs, physical exam, and clinical laboratory assessments.

SECONDARY OUTCOMES:
Overall response according to RECIST guidelines (version 1.1, 2009) | Computed tomography (CT) scans for tumor imaging will be performed at the end of every 2 treatment cycles (8 weeks) and an average of 4 cycles (16 weeks)
  The determination of antitumor efficacy will be based on objective tumor assessments made by the investigator according to RECIST guidelines (version 1.1, 2009).

OTHER OUTCOMES:
Area under the concentration time curve (AUC) | During Dose Escalation Phase PK blood samples for determination of TAS-119 PK profile will be collected during Cycle 1. In the Expansion Phase, the first 12 patients (DDI Subgroup) will undergo PK sampling in Cycle 1 and Cycle 2 (up to 31 days).
  During Dose Escalation Phase PK blood samples will be collected from each arm during Cycle 1 (predose up to 24 hours post-dose). In the Expansion Phase, the first 12 patients (DDI Subgroup) of each arm will undergo PK sampling in Cycle 1 (predose up to 24 hours) and Cycle 2 (predose up to 48 hours post-dose).
Maximum Plasma Concentration (Cmax) | During Dose Escalation Phase PK blood samples for determination of TAS-119 PK profile will be collected during Cycle 1. In the Expansion Phase, the first 12 patients (DDI Subgroup) will undergo PK sampling in Cycle 1 and Cycle 2 (up to 31 days).
  During Dose Escalation Phase PK blood samples will be collected from each arm during Cycle 1 (predose up to 24 hours post-dose). In the Expansion Phase, the first 12 patients (DDI Subgroup) of each arm will undergo PK sampling in Cycle 1 (predose up to 24 hours) and Cycle 2 (predose up to 48 hours post-dose).
Time of maximum observed serum concentration (Tmax) | During Dose Escalation Phase PK blood samples for determination of TAS-119 PK profile will be collected during Cycle 1. In the Expansion Phase, the first 12 patients (DDI Subgroup) will undergo PK sampling in Cycle 1 and Cycle 2 (up to 31 days).
  During Dose Escalation Phase PK blood samples will be collected from each arm during Cycle 1 (predose up to 24 hours post-dose). In the Expansion Phase, the first 12 patients (DDI Subgroup) of each arm will undergo PK sampling in Cycle 1 (predose up to 24 hours) and Cycle 2 (predose up to 48 hours post-dose).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Colorado Hospital Anschutz Cancer Pavilion, Aurora, Colorado
  - Washington University School of Medicine Division of Oncology Siteman Cancer Center, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee